CLINICAL TRIAL: NCT04032756
Title: Tofacitinib Registry of Patients With Ulcerative Colitis in Germany - Documentation of Tofacitinib Induction and Maintenance Therapy in Conjunction With Long-term Outcome and Predictors of Response
Brief Title: Tofacitinib Registry of Patients With Ulcerative Colitis in Germany
Acronym: TOFA-UC
Status: Terminated | Type: Observational
Why Stopped: not enough patients recruited, Study objective could not be achieved
Sponsor: Ced Service GmbH (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: Protocol V1.4 31.05.2019
Record Dates: First submitted 2019-07-19; First posted 2019-07-25 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Colitis, Ulcerative; Biologics; Tofacitiniib; Chronic Inflammatory Small Bowel Disease; Bowel Diseases, Inflammatory; Bowel Disease; CED
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases; Intestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: UC-patients (age at enrollment: 18-80 years) receiving a newly introduced Tofacitinib therapy (n=360). Previous treatment(s) with biologics or immunosuppressants is (are) permitted. About 20-30% of the Tofacitinib patients will biologic-naiv.
- Group 2: UC-patients (age at enrollment: 18-80 years) receiving a newly introduced biologics therapy (n=120). Previous treatment(s) with biologics or immunosuppressants is (are) allowed.

SUMMARY:
This registry on Tofacitinib and biologics (anti-integrin/anti-TNF) in the treatment of ulcerative colitis (UC) patients in Germany will extend the prospective documentation of safety issues and efficacy in induction and maintenance therapy of Tofacitinib (Xeljanz®) in addition to other biologics used in Germany with a particular interest in predictors of long-term responses and favorable disease outcome or to predict severe side effects caused by therapy with Januskinase(JAK)- inhibitors/biologics.

DETAILED DESCRIPTION:
This is an Investigator-initiated non-randomized, non-interventional observational prospective long- term research (IIR) as part of the normal treatment of UC patients for the safety and efficacy of Tofacitinib / biologic therapies. As of 01st July 2019, UC patients who have been provided Tofacitinib / biologics for UC according the respective label by the treating physician may be prospectively included in an online database by the participating study centers by 31st March 2021.

An interim analysis is planned at the end of patients ́ recruitment with respect of the induction phase (week 16) for October 2021 with a first publication of the data in a peer-reviewed journal (e.g., JCC, GUT, UEG Journal).

Up to 480 patients (including about 360 UC patients with Tofacitinib and about 120 UC patients with biologics) will be included in the online documentation. A specification to the study centers regarding the group inclusion (patients treated with Tofacitinib (group 1) or a biologics (group 2)) will not be made; this means, each study center can include patients in both groups.

The CED Service GmbH assume that approximately 20-30% of Tofacitinib patients will be biologic-naïve UC patients, many of whom will represent early disease patients (< 2 years after first diagnosis).

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe Ulcerative Colitis aged 18-80 years at enrollment
* Written informed consent is given

Exclusion Criteria:

* Malignant disease in history (except for non-melanoma skin cancer)
* Any contraindication according to the SmPC of the respective medication

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Up to 480 patients (aged 18-80 years at enrollment) (including about 360 UC patients with Tofacitinib and about 120 UC patients with biologics) will be included in the online documentation. A specification to the study centers regarding the group inclusion (patients treated with Tofacitinib (group 1) or a biologics (group 2)) will not be made; this means, each study center can include patients in both groups.
  The CED Service GmbH assume that approximately 20-30% of Tofacitinib patients will be biologic-naïve UC patients, many of whom will represent early disease patients (< 2 years after first diagnosis).
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
partial Mayo score ≤ 1 plus a bleeding subscore of 0) in the inductionphase (week 16) | 07/01/2019 - 03/31/2023
  The primary endpoint is steroid-free remission (remission: partial Mayo score ≤ 1 plus a bleeding subscore of 0) in the inductionphase (week 16). For this endpoint it will be only captured if there is a current use of steroids at the time of the visit. So the patient will be asked for current steroid use at time of visit at week 16 and if he has received steroids within the last 4 weeks prior to time point of the visit.

SECONDARY OUTCOMES:
occurrence of serious side effects (e.g., death, tumor, tuberculosis, severe infections, or side effects leading to hospitalization) | 07/01/2019 - 03/31/2023
  Online documentation of safety and efficacy in induction and maintenance therapy including the occurrence of serious side effects (e.g., death, tumor, tuberculosis, severe infections, or side effects leading to hospitalization)
response: partial Mayo Score reduction of ≥ 3 accompanied by a decrease of at least 30% from baseline and remission: partial Mayo score ≤ 1 plus a bleeding subscore of 0 - Efficacy | 07/01/2019 - 03/31/2023
  Efficacy (response: partial Mayo Score reduction of ≥ 3 accompanied by a decrease of at least 30% from baseline and remission: partial Mayo score ≤ 1 plus a bleeding subscore of 0) of induction therapy (week 8 and 16) and maintenance therapy (months 6 to 24) and efficacy (response and remission) in different subpopulations, e.g. based on a previous biologic therapy or not.
hospitalization days via question in questionnaire | 07/01/2019 - 03/31/2023
  Obtaining health economic data in UC patients on Tofacitinib / biologics therapy (hospitalization)
psychosocial impairments - EQ-5D | 07/01/2019 - 03/31/2023
  Obtaining data of the course from UC patients with a new therapy (Tofacitinib / biologics) related to treatment strategy and psychosocial impairments
EQ-5D quality of life | 07/01/2019 - 03/31/2023
  Obtaining health economic data in UC patients on Tofacitinib / biologics therapy (quality of life)
early retirement via question in questionnaire | 07/01/2019 - 03/31/2023
  Obtaining health economic data in UC patients on Tofacitinib / biologics therapy (early retirement)

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterologische Gemeinschaftspraxis Minden, Minden, Lower Saxony, Germany

DOCUMENTS (1):
  • Study Protocol (2019-05-31): https://cdn.clinicaltrials.gov/large-docs/56/NCT04032756/Prot_000.pdf